CLINICAL TRIAL: NCT01445652
Title: A Lifestyle Investigation With Spectacles and Daily Disposable Contact Lenses in Young Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-370-C-091 / CB11-500
Record Dates: First submitted 2011-09-30; First posted 2011-10-04 (Estimated); Results first posted 2013-09-09 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Eyeglasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nelfilcon A (Experimental): Nelfilcon A contact lenses worn in both eyes on a daily disposable basis a minimum of five days per week, eight hours per day, for six months
  Interventions: Device: nelfilcon A contact lens
- Spectacles (Active Comparator): Spectacles per current prescription worn a minimum of five days per week, eight hours per day, for six months
  Interventions: Other: Spectacles

INTERVENTIONS:
Device: nelfilcon A contact lens — Commercially marketed, single vision, soft contact lens for daily disposable wear
  Other Names: DAILIES AQUACOMFORT PLUS
  Arms: nelfilcon A
Other: Spectacles — Spectacles per current prescription
  Arms: Spectacles

SUMMARY:
The purpose of this study was to evaluate the relative benefits of daily disposable contact lenses versus spectacles in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Understands rights as a research subject and willing and able to sign a Statement of Informed Consent, or if under 18, parent or guardian understands rights and is willing and able to sign a Statement of Informed Consent.
* Willing and able to follow the protocol.
* Currently wearing spectacles full-time (at least five days per week, eight hours per day).
* Has never worn contact lenses (more than one day) before.
* Agrees to not participate in other clinical research for the duration of this study.
* Can attain at least 6/9 in each eye with the study optical correction.
* Can be fitted with study lenses in the available power range (contact lens group) or can select a satisfactory spectacle lens frame and lenses (spectacle group).
* Willing and able to wear the study lenses or spectacles for a minimum of five days per week, eight hours per day.
* Owns or has regular access to a mobile phone and is familiar with SMS text messaging.
* Has an up-to-date and functional pair of spectacles at time of enrollment.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Has an ocular or systemic disorder that would normally contraindicate contact lens wear.
* Is using any topical medication such as eye drops or ointment.
* Has had corneal refractive surgery.
* Has had cataract surgery.
* Has diabetes.
* Has taken part in other clinical research within two weeks of starting the study.
* Other protocol-defined exclusion criteria may apply.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 113 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, PhD MCOptom FAAO FBCLA, Principal Investigator — University of Manchester
Locations (1):
- Eurolens Research, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from one study center in the United Kingdom.
Pre-assignment Details: Of the 113 participants enrolled, 3 were exited as screen failures prior to randomization. This reporting group includes all enrolled and randomized participants (110).
Period: Overall Study
Arm/Group | Nelfilcon A | Spectacles
Started | 57 | 53
Completed | 47 | 50
Not Completed | 10 | 3
Not completed — Not comfortable in lenses | 5 | 0
Not completed — Failed to attend scheduled visit | 2 | 3
Not completed — Failed teach session | 2 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: This reporting group includes all enrolled and randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nelfilcon A | Spectacles | Total
Number analyzed (Participants) | 57 | 53 | 110
Age Continuous [Mean (Standard Deviation); unit: years] | 16.2 (1.8) | 16.3 (2.0) | 16.2 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 25 | 22 | 47
Region of Enrollment [Number; unit: participants]
  United Kingdom | 57 | 53 | 110

OUTCOME MEASURES:

1. Primary Outcome: Subjective Happiness With Correction Type
Description: Participant responded to an SMS message: "Please rate your happiness (H) and vision (V) with your [contact lenses/spectacles]: 1=very poor; 2=poor; 3=neither; 4=good; and 5=very good. eg H2V4. Please send N if in you are not wearing [contact lenses/spectacles]."
Time Frame: Month 6
Population: This reporting group includes all participants who sent in an SMS response.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Nelfilcon A | Spectacles
Number analyzed (Participants) | 14 | 21
Units on a Scale | 4.92 (0.3) | 4.50 (0.9)

2. Primary Outcome: Subjective Vision With Correction Type
Description: as for outcome 1
Time Frame: Month 6
Population: This reporting group includes all participants who sent in an SMS response.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nelfilcon A | Spectacles
Number analyzed (Participants) | 14 | 21
Units on a scale | 4.5 (0.7) | 4.5 (0.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (9 months). An adverse event was defined as any unfavourable or unintended sign or symptom associated with the use of a contact lens, but not necessarily caused by the contact lens.
Description: This reporting group includes all enrolled and randomized participants.
Arm/Group | Nelfilcon A | Spectacles
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/53
Other Adverse Events (participants affected / at risk) | 4/57 | 0/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nelfilcon A (N=57) | Spectacles (N=53)
Corneal inflammatory event (Eye disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.